CLINICAL TRIAL: NCT00987844
Title: A Study to Evaluate the Long-Term Tolerability, Safety, Patient Satisfaction, Pharmacokinetics, and Use Patterns of Oral Prucalopride Tablets in Patients With Chronic Constipation
Brief Title: Study to Evaluate Long-Term Safety, Tolerability, and Satisfaction With Prucalopride in Chronic Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Movetis (Industry)
Responsible Party: Renate Specht Gryp, Movetis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRU-USA-22
Record Dates: First submitted 2009-09-24; First posted 2009-10-01 (Estimated); Last update posted 2009-10-01 (Estimated); Status verified 2009-09

CONDITIONS: Chronic Constipation
MeSH Terms: interventions — prucalopride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Prucalopride — 1 mg tablets, free dosing regiment with max. of 4 tablets o.d., treatment duration: up to 24 months

SUMMARY:
Objectives: To evaluate the clinical long-term safety and the tolerability, patient satisfaction, pharmacokinetics and use of pattern of prucalopride given in doses up to 4 mg per day to patients with chronic constipation (CC).

ELIGIBILITY:
Inclusion Criteria:

1. Male and non-pregnant, non breast-feeding female outpatients at least 18 years of age.
2. Patient completed the entire treatment period of one of the following studies: PRU-USA-3, PRU-USA-11, PRU-USA-13, PRU-USA-21, PRU-USA-25, PRU-USA-27 or PRU-USA-28, or Patient participated in the re-treatment study PRU-USA-28 and did not qualify for Treatment period II after both washout periods.

Exclusion Criteria:

1. Patient with impaired renal function
2. Patient with clinically significant abnormalities of haematology, urinalysis, or blood chemistry.
3. Female of childbearing potential without adequate contraceptive protection during the study.
4. Patient who used an investigation drug other than prucalopride in the 30 days preceding the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1775 (Actual)
Dates: Start 1998-07; Primary Completion 2000-11 (Actual)

PRIMARY OUTCOMES:
Safety: adverse events, lab tests, vital signs, ECGs | 24 months

SECONDARY OUTCOMES:
Efficacy: PAC-QOL self-administered questionnaire, Patient's pattern of use of prucalopride | 24 months
Pharmacokinetics: Prucalopride plasmaconcentrations | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Camilleri M, Van Outryve MJ, Beyens G, Kerstens R, Robinson P, Vandeplassche L. Clinical trial: the efficacy of open-label prucalopride treatment in patients with chronic constipation - follow-up of patients from the pivotal studies. Aliment Pharmacol Ther. 2010 Nov;32(9):1113-23. doi: 10.1111/j.1365-2036.2010.04455.x. Epub 2010 Sep 16. PMID 21039673